CLINICAL TRIAL: NCT03836872
Title: Acupuncture for Joint Symptoms in Patients With Breast Cancer: A Randomised Controlled Trial
Brief Title: Acupuncture for Joint Symptoms in Patients With Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: China has experienced new waves of COVID-19 since January 2021, and the Chinese government has adopted strict COVID-19 policies to control the occasional outbreaks of COVID-19.
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The Affiliated Hospital Of Southwest Medical University (Other)
Responsible Party: Principal Investigator, Professor Alex MOLASIOTIS, Chair Professor of Nursing and Head, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20180509004
Record Dates: First submitted 2019-02-01; First posted 2019-02-11 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Female Breast Cancer
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- True Acupuncture (Experimental): Patients in the experimental group will receive, in addition to standard care, a standardised 30-minute acupuncture session needling specific acupoints. Bilateral acupoints will be stimulated including Waiguan (SJ5), Jianjing (GB21), Yanglingquan (GB34), Hegu (LI4), Jiexi (ST41) and Taixi (K3). In addition, joint specific acupoints will also be used, depending on where the joint symptoms are present.
  Interventions: Device: Acupuncture
- Sham Acupuncture (Sham Comparator): In addition to the routine methods of care, patients allocated to the sham control group will receive sham acupuncture treatment at sham acupoints with superficial needling
  Interventions: Device: Acupuncture
- Standard Control Group (No Intervention): The third arm will be a standard care control arm.

INTERVENTIONS:
Device: Acupuncture — Patients in the experimental group will receive, in addition to standard care, a standardised 30-minute acupuncture session needling specific acupoints although there will be flexibility in case some points cannot be punctured (e. g. in case of lymphoedema), and alternative points (as in routine practice) may be selected by the acupuncture practitioner using their discretion to maintain an equal dose of treatment to all patients. Bilateral acupoints will be stimulated. These points will include Waiguan (SJ5), Jianjing (GB21), Yanglingquan (GB34), Hegu (LI4), Jiexi (ST41) and Taixi (K3). In addition, joint specific acupoints will also be used, depending on where the joint symptoms are present.
  Arms: Sham Acupuncture; True Acupuncture

SUMMARY:
Joint symptoms including stiffness, local pain and aches are common adverse reactions among breast cancer (BC) patients undergoing hormone treatments, while effective interventions for managing such symptoms have not been well explored so far. Acupuncture can be a promising approach to controlling joint symptoms in BC patients but current research evidence generated from several small-scale clinical studies have not been robust enough to support the use of acupuncture for cancer symptom management in routine practice.

The overall aim of the research project is to examine the effectiveness of a 6-week acupuncture protocol for the management of joint symptoms in Chinese female BC patients who are currently undergoing hormone treatments following the completion of taxane-based chemotherapy. Given the lack of available data regarding the prevalence of joint symptoms in BC patients in mainland China, a large cross-sectional survey will also be performed to examine the incidence of joint symptoms among Chinese BC patients in mainland China and the impact of joint symptoms on patients' quality of life.

DETAILED DESCRIPTION:
A three-group trial design is proposed, with an experimental group receiving true acupuncture at specific acupuncture points, a sham control group receiving sham acupuncture at non-acupuncture Acupoints with superficial needling, both in addition to routine methods of care, and a group receiving usual care only.

Participants and Settings BC patients who have completed taxane-based chemotherapy and are currently receiving hormone treatments with the experience of joint pain will be the targeted study population. The study will take place in the Southwest Medical University Hospital, a large medical centre in Sichuan, China.

Sample Size 55 per group (165 in total).

The Intervention Protocol

1. True Acupuncture Protocol will be used in the True Acupuncture Group (Experimental Group)

   The acupuncture intervention is described below based on the STRICTA recommendations for reporting acupuncture trials. Patients in the experimental group will receive, in addition to standard care, a standardised 30-minute acupuncture session needling specific acupoints although there will be flexibility in case some points cannot be punctured (e. g. in case of lymphoedema), and alternative points (as in routine practice) may be selected by the acupuncture practitioner using their discretion to maintain an equal dose of treatment to all patients. Bilateral acupoints will be stimulated. These points will include Waiguan (SJ5), Jianjing (GB21), Yanglingquan (GB34), Hegu (LI4), Jiexi (ST41) and Taixi (K3). In addition, joint specific acupoints will also be used, depending on where the joint symptoms are present. The additional acupoints will be:
   1. Shoulder (Bilateral Acupoints): Jianyu (LI15), Jianliao (SJ14), and Naoshu (SI10); The following alternative acupoints would be considered in case of some patients may have lymphoedema or other problem at particular sites where the above proposed acupoints cannot be stimulated: Quchi (LI11), Shousanli (LI10), Tianzong (SI11) and Taichong (LR3).
   2. Wrist (Bilateral Acupoints): Yangchi (SJ4), Yangxi (LI5), and Daling (PC7); The following alternative acupoints would be considered in case of some patients may have lymphoedema or other problem at particular sites where the above proposed acupoints cannot be stimulated: Zhigou (SJ6), Jianshi (PC5) and Wailaogong (EX-UE8).
   3. Fingers (Bilateral Acupoints): Yanggu (SI5), Houxi (SI3), and Sanjian (LI3); Alternative acupoints located on the wrist or forearm would be considered in case of some patients may have lymphoedema or other problem at particular sites where the above proposed acupoints cannot be stimulated.
   4. Lumbar Area (Bilateral Acupoints): Yaoyangguan (DU3), Jingsuo (DU8), and Shenyu (BL23); Alternative acupoint Weizhong (BL40) located on the wrist or forearm would be considered in case of some patients may have lymphoedema or other problem at particular sites where the above proposed acupoints cannot be stimulated.
   5. Hip (Bilateral Acupoints): Huantiao (GB30), Xuanzhong (GB39), and Juliao (GB29); The following alternative acupoints would be considered in case of some patients may have lymphoedema or other problem at particular sites where the above proposed acupoints cannot be stimulated: Fengshi (GB31) and Biguan (ST31).
   6. Knee (Bilateral Acupoints): Yinlingquan (SP9), Xuehai (SP10), and Liangqiu (ST34).

   The following alternative acupoints would be considered in case of some patients may have lymphoedema or other problem at particular sites where the above proposed acupoints cannot be stimulated: Heding (EX-LE2), Futu (ST32), Baichongwo (EX-LE3), and Xiyan (EX-LE5).

   Acupuncture will be twice a week for consecutive 6 weeks, thus a total of 12 sessions of acupuncture will be carried out.
2. Sham Acupuncture Protocol will be used in the Sham Acupuncture Group (Sham Control Group) In addition to the routine methods of care, patients allocated to the sham control group will receive sham acupuncture treatment at sham acupoints with superficial needling to avoid the generation of specific treatment effects. The sham acupoints selected for stimulation will be those located 1-3 cm near the true acupoints used in the true acupuncture group. The number of the selected sham acupoints will be the same as those used in the true acupuncture group. Meanwhile, to maintain the homogeneity of the routine methods of care used across groups, the conventional care for all the participants in this study will include at least written education materials in terms of the knowledge of joint symptoms and instructions of the use of painkillers and non-steroidal anti-inflammatory drugs (NSAIDs). During the whole study period, the study investigators will also record any other treatments, including other complementary and alternative approaches, that participants may receive and view as potential confounders in the data analysis stage. Given the design of true and sham acupuncture groups, participants, study investigators and outcome assessors will not know the actual group assignment of the true and sham acupuncture group, and a partial blinding design is therefore utilized for this proposed study.
3. Usual care wil be used in the waiting-list control group (Waiting-list Control Group) Participants in this group will only receive the usual care for the period that they are on the waiting list. But the waiting-list control group will offer acupuncture intervention after the completion of the RCT.

Study Duration and Outcome Assessment The total acupuncture treatment duration will be six weeks, and the duration of study involvement for each participant will be around 20 weeks including baseline assessment, immediate post-treatment assessment after the 6-week acupuncture, and two follow-up assessment at 12 weeks and 20 weeks, respectively.

Ethical Considerations A written informed consent will be obtained from every eligible person agreeing to participate after the risks and benefits of the study have been explained to them verbally and in writing. Participation in the study is on a voluntary basis, and all potential participants will be informed and assured that they have the right to refuse or withdraw from the study at any time. Personal information and data will remain confidential and anonymous. Side effects arising from acupuncture are rare. However, abnormal phenomena such as local tenderness, fainting, stuck needle, bent needle, broken needle, and haematoma during or after the procedure may be possible. Such conditions will be resolved quickly when the needles are removed, and the client's conditions will be monitored closely and recorded. Application for ethical approval from the Human Research Ethics Review Committee has been obtained from The Hong Kong Polytechnic University and the hospital where the trial will be carried out.

Data Analysis Analyses will include descriptive statistics to summarise the data, analysis of variance to assess between-groups differences, and regression analysis (such as ANCOVA) using the baseline pain score as covariate. 95% CIs will also be calculated. In more detail, while a t-test is adequate for analysis, analysis of covariance will be used with the baseline pain score as a covariate and centre and trial arm as grouping factors. Equivalent analyses will be performed for the week 20 data (although it is acknowledged that such analyses would not be independent of the 12-week scores, as it is likely the week-12 and week-20 values will be correlated). Drop-out cases and non-respondents will be asked to complete 1 item about their pain levels from the BPI scale to capture outcomes in as many patients as possible in the intention to treat analysis.

Significance and Implications Using robust methodology the study will investigate and interpret the use, delivery and outcomes of acupuncture in the management of a debilitating symptom of cancer therapies in order to inform decision-making and policy-making, and contribute to the evidence base for the treatment of hormone treatment-related joint symptoms. This study will provide information that can lead to improvements in the care of cancer patients, have a positive impact on quality of life and may increase the number of patients successfully completing hormone treatments. The project is about complementary therapies that many cancer patients frequently use, and has the potential to translate into benefits for patients fairly quickly. An information booklet on managing joint pains in breast cancer patients would also be a key outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

1. BC patients with a confirmed diagnosis of hormone receptor-positive BC at the stage of I, II or IIIa;
2. Patients who have completed taxane-based chemotherapy and are currently undergoing hormone treatments for at least three months;
3. Patients indicate ongoing joint symptoms, including joint pain and/or stiffness, at one or more sites of body;
4. Patients started to experience the joint symptoms after the commencement of the hormone treatments;
5. Patients indicate the intensity of their worst pain during the past seven days of greater than 4 points at a 0-10 NRS scale where 0 represents no pain and 10 indicates most severe pain;
6. Patients have at least a primary school education and are able to communicate in Chinese Mandarin or Sichuanese; and
7. Patients agree to participate in the trial and are willing to give written informed consent.

Exclusion Criteria:

1. Patients who had needle phobia and a low count of platelet of less than 50,000;
2. Patients with conditions which are not appropriate for acupuncture including pregnancy, bleeding disorders, local or systematic inflammation, and other neuropathic and/or metabolic problems of the joints;
3. Patients who had received joint surgery or had bone fracture during the past six months;
4. Patients who had received any types of acupoint stimulation (e.g. body acupuncture or acupressure and auricular therapy) during the past six months; and
5. Patients are currently treated with narcotic analgesia or steroids.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory | 6-week assessment
  Pain assessment measuring intensity of pain and impact of pain on daily functions. All items on a 0-10 numerical rating scale. Higher scores indicate worse pain and worse impact in daily lives.

SECONDARY OUTCOMES:
Manchester Foot Pain Disability Questionnaire | 6-week assessment
  Measures foot pain with 19 items and three dimensions (functioning limitations with 12 items; pain intensity with 4 items; personal appearance with 3 items). Higher scores indicate worse outcomes.
Manchester Foot Pain Disability Questionnaire | 12-week assessment
  Measures foot pain with 19 items and three dimensions (functioning limitations with 12 items; pain intensity with 4 items; personal appearance with 3 items). Higher scores indicate worse outcomes.
Manchester Foot Pain Disability Questionnaire | 20-week assessment
  Measures foot pain with 19 items and three dimensions (functioning limitations with 12 items; pain intensity with 4 items; personal appearance with 3 items). Higher scores indicate worse outcomes.
Michigan Hand Outcomes Questionnaire | 6-week assessment
  Assesses hand function with 37 items, and has 6 dimensions of hand functioning
Michigan Hand Outcomes Questionnaire | 12-week assessment
  Assesses hand function with 37 items, and has 6 dimensions of hand functioning
Michigan Hand Outcomes Questionnaire | 20-week assessment
  Assesses hand function with 37 items, and has 6 dimensions of hand functioning
Western Ontario & McMaster Universities Osteoarthritis Index | 6-week assessment
  Assesses 3 dimensions of osteoarthritis symptoms with 24 items, including joint pain, stiffness and disability. Higher scores are indicative of worse functioning and higher symptom burden.
Western Ontario & McMaster Universities Osteoarthritis Index | 12-week assessment
  Assesses 3 dimensions of osteoarthritis symptoms with 24 items, including joint pain, stiffness and disability. Higher scores are indicative of worse functioning and higher symptom burden.
Western Ontario & McMaster Universities Osteoarthritis Index | 20-week assessment
  Assesses 3 dimensions of osteoarthritis symptoms with 24 items, including joint pain, stiffness and disability. Higher scores are indicative of worse functioning and higher symptom burden.
Arthritis Impact Measurement Scale 2-Short Form | 6-week assessment
  Assesses arthritis-related quality of life with 26 items in 5 domains (physical functioning, symptoms, impact, social and functional dimensions), with higher scores indicating worse quality of life.
Arthritis Impact Measurement Scale 2-Short Form | 12-week assessment
  Assesses arthritis-related quality of life with 26 items in 5 domains (physical functioning, symptoms, impact, social and functional dimensions), with higher scores indicating worse quality of life.
Arthritis Impact Measurement Scale 2-Short Form | 20-week assessment
  Assesses arthritis-related quality of life with 26 items in 5 domains (physical functioning, symptoms, impact, social and functional dimensions), with higher scores indicating worse quality of life.
Functional Assessment of Cancer Therapy-Breast | 6-week assessment
  This is a disease specific quality of life assessment scale. Higher scores indicate better quality of life outcomes.
Functional Assessment of Cancer Therapy-Breast | 12-week assessment
  This is a disease specific quality of life assessment scale. Higher scores indicate better quality of life outcomes.
Functional Assessment of Cancer Therapy-Breast | 20-week assessment
  This is a disease specific quality of life assessment scale. Higher scores indicate better quality of life outcomes.
Medical Outcomes Survey 36-item short form version | 6-week assessment
  It measures quality of life with 36 items assessing eight health concepts, including bodily pain, role limitations and emotional well-being. Higher scores indicate worse quality of life outcomes.
Medical Outcomes Survey 36-item short form version | 12-week assessment
  It measures quality of life with 36 items assessing eight health concepts, including bodily pain, role limitations and emotional well-being. Higher scores indicate worse quality of life outcomes.
Medical Outcomes Survey 36-item short form version | 20-week assessment
  It measures quality of life with 36 items assessing eight health concepts, including bodily pain, role limitations and emotional well-being. Higher scores indicate worse quality of life outcomes.
Brief Pain Inventory | 12 weeks assessment
  Brief Pain Inventory (BPI) measuring intensity of pain and impact of pain on daily functions. All items on a 0-10 numerical rating scale. Higher scores indicate worse pain and worse impact in daily lives.
Brief Pain Inventory | 20 weeks assessment
  Brief Pain Inventory (BPI) measuring intensity of pain and impact of pain on daily functions. All items on a 0-10 numerical rating scale. Higher scores indicate worse pain and worse impact in daily lives.

OTHER OUTCOMES:
Questionnaire for Patient Sociodemographic and Clinical Characteristics | baseline assessment
  Sample characteristics obtained in a descriptive manner (i.e. sex; education level, stage of disease; duration of hormone treatment etc).

CONTACTS AND LOCATIONS:
Overall Officials: Alex Molassiotis, PhD, Study Chair — The Hong Kong Polytechnic University
Locations (1):
- Xianliang Liu, Luzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cleeland, C.S., Pain assessment in cancer. In: D. Osoba (Ed.), Effect of Cancer on Quality of Life, CRC Press, Boca Raton, FL, 1991, 293-305.
- [Background] Cleeland, C. S. (2014). The brief pain inventory user guide. 2009. Cleeland Charles S, Houston, TX Google Scholar.
- [Background] Wang XS, Mendoza TR, Gao SZ, Cleeland CS. The Chinese version of the Brief Pain Inventory (BPI-C): its development and use in a study of cancer pain. Pain. 1996 Oct;67(2-3):407-16. doi: 10.1016/0304-3959(96)03147-8. PMID 8951936
- [Background] Brady MJ, Cella DF, Mo F, Bonomi AE, Tulsky DS, Lloyd SR, Deasy S, Cobleigh M, Shiomoto G. Reliability and validity of the Functional Assessment of Cancer Therapy-Breast quality-of-life instrument. J Clin Oncol. 1997 Mar;15(3):974-86. doi: 10.1200/JCO.1997.15.3.974. PMID 9060536
- [Background] Chung KC, Pillsbury MS, Walters MR, Hayward RA. Reliability and validity testing of the Michigan Hand Outcomes Questionnaire. J Hand Surg Am. 1998 Jul;23(4):575-87. doi: 10.1016/S0363-5023(98)80042-7. PMID 9708370
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Crew KD, Capodice JL, Greenlee H, Apollo A, Jacobson JS, Raptis G, Blozie K, Sierra A, Hershman DL. Pilot study of acupuncture for the treatment of joint symptoms related to adjuvant aromatase inhibitor therapy in postmenopausal breast cancer patients. J Cancer Surviv. 2007 Dec;1(4):283-91. doi: 10.1007/s11764-007-0034-x. Epub 2007 Oct 12. PMID 18648963
- [Background] Crew KD, Capodice JL, Greenlee H, Brafman L, Fuentes D, Awad D, Yann Tsai W, Hershman DL. Randomized, blinded, sham-controlled trial of acupuncture for the management of aromatase inhibitor-associated joint symptoms in women with early-stage breast cancer. J Clin Oncol. 2010 Mar 1;28(7):1154-60. doi: 10.1200/JCO.2009.23.4708. Epub 2010 Jan 25. PMID 20100963
- [Background] Crew KD, Greenlee H, Capodice J, Raptis G, Brafman L, Fuentes D, Sierra A, Hershman DL. Prevalence of joint symptoms in postmenopausal women taking aromatase inhibitors for early-stage breast cancer. J Clin Oncol. 2007 Sep 1;25(25):3877-83. doi: 10.1200/JCO.2007.10.7573. PMID 17761973
- [Background] de Barros EN, Alexandre NM. Cross-cultural adaptation of the Nordic musculoskeletal questionnaire. Int Nurs Rev. 2003 Jun;50(2):101-8. doi: 10.1046/j.1466-7657.2003.00188.x. PMID 12752909
- [Background] Dawson J, Fitzpatrick R, Murray D, Carr A. Questionnaire on the perceptions of patients about total knee replacement. J Bone Joint Surg Br. 1998 Jan;80(1):63-9. doi: 10.1302/0301-620x.80b1.7859. PMID 9460955
- [Background] Dunbar MJ, Robertsson O, Ryd L, Lidgren L. Translation and validation of the Oxford-12 item knee score for use in Sweden. Acta Orthop Scand. 2000 Jun;71(3):268-74. doi: 10.1080/000164700317411861. PMID 10919298
- [Background] Fan CY, Jiang J, Zeng BF, Jiang PZ, Cai PH, Chung KC. Reconstruction of thumb loss complicated by skin defects in the thumb-index web space by combined transplantation of free tissues. J Hand Surg Am. 2006 Feb;31(2):236-41. doi: 10.1016/j.jhsa.2005.10.021. PMID 16473684
- [Background] Li L, Wang H, Shen Y. Development and psychometric tests of a Chinese version of the SF-36 Health Survey Scales. Zhonghua Yu Fang Yi Xue Za Zhi. 2002 Mar;36(2):109-13. PMID 12410965
- [Background] Hill J, Bird HA, Lawton CW, Wright V. The arthritis impact measurement scales: an anglicized version to assess the outcome of British patients with rheumatoid arthritis. Br J Rheumatol. 1990 Jun;29(3):193-6. doi: 10.1093/rheumatology/29.3.193. PMID 2357501
- [Background] Manheimer E, Cheng K, Linde K, Lao L, Yoo J, Wieland S, van der Windt DA, Berman BM, Bouter LM. Acupuncture for peripheral joint osteoarthritis. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD001977. doi: 10.1002/14651858.CD001977.pub2. PMID 20091527
- [Background] Ostendorf M, van Stel HF, Buskens E, Schrijvers AJ, Marting LN, Verbout AJ, Dhert WJ. Patient-reported outcome in total hip replacement. A comparison of five instruments of health status. J Bone Joint Surg Br. 2004 Aug;86(6):801-8. doi: 10.1302/0301-620x.86b6.14950. PMID 15330018
- [Background] Wan C, Zhang D, Yang Z, Tu X, Tang W, Feng C, Wang H, Tang X. Validation of the simplified Chinese version of the FACT-B for measuring quality of life for patients with breast cancer. Breast Cancer Res Treat. 2007 Dec;106(3):413-8. doi: 10.1007/s10549-007-9511-1. Epub 2007 Mar 22. PMID 17377841
- [Background] Xie F, Li SC, Lo NN, Yeo SJ, Yang KY, Yeo W, Chong HC, Fong KY, Thumboo J. Cross-cultural adaptation and validation of Singapore English and Chinese Versions of the Oxford Knee Score (OKS) in knee osteoarthritis patients undergoing total knee replacement. Osteoarthritis Cartilage. 2007 Sep;15(9):1019-24. doi: 10.1016/j.joca.2007.02.013. Epub 2007 Apr 3. PMID 17408984
- [Background] Zhu, J., Zhang, Y., Pang, L., & Fu, H. (2006) Test of Reliability and Validity of Short-Form Arthritis Impact Measurement Scales2 (AIMS2-SF). Chinese Journal of Prevention and Control of Chronic Non- Communicable Diseases, 14: 7577.